CLINICAL TRIAL: NCT03931538
Title: Urinary Tract Infection: RapID Molecular Organism Identification and Mixed Flora Antibiotic Resistance Profiling (MixAR)
Brief Title: Rapid Molecular Organism Identification and Mixed Flora Antibiotic Resistance Profiling (MixAR) Prospective Study
Acronym: RapIDMixAR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pathnostics (Industry)
Collaborators: Comprehensive Urology-a Division of Michigan Healthcare Professionals (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Diagnostic
Other Study IDs: Pathnostics RapID MixAR
Record Dates: First submitted 2019-04-25; First posted 2019-04-30 (Actual); Last update posted 2023-08-28 (Actual); Status verified 2023-08

CONDITIONS: Urinary Tract Infections; Prostatitis; Interstitial Cystitis
Keywords: UTI; IC
MeSH Terms: conditions — Urinary Tract Infections; Prostatitis; Cystitis, Interstitial

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Culture Only (Active Comparator): Physician receives only culture result
  Interventions: Diagnostic Test: Urine Culture
- Guidance 4.0 PCR test only (Active Comparator): Physician receives Guidance report only
  Interventions: Diagnostic Test: Guidance 4.0 PCR test
- Culture and Guidance 4.0 PCR test Group (Active Comparator): Physician receives both results, gets Culture report immediately before Guidance
  Interventions: Diagnostic Test: Guidance 4.0 PCR test; Diagnostic Test: Urine Culture
- Guidance 4.0 PCR test and culture group (Active Comparator): Physician receives both results, gets Guidance report immediately before culture
  Interventions: Diagnostic Test: Guidance 4.0 PCR test; Diagnostic Test: Urine Culture

INTERVENTIONS:
Diagnostic Test: Guidance 4.0 PCR test — All patients will have a urine culture and Guidance 4.0 PCR test run on their urine, but physicians will receive one or the other, or both depending on the treatment arm.
  Arms: Culture and Guidance 4.0 PCR test Group; Guidance 4.0 PCR test and culture group; Guidance 4.0 PCR test only
Diagnostic Test: Urine Culture — All patients will have a urine culture and Guidance 4.0 PCR test run on their urine, but physicians will receive one or the other, or both depending on the treatment arm.
  Arms: Culture Only; Culture and Guidance 4.0 PCR test Group; Guidance 4.0 PCR test and culture group

SUMMARY:
In this protocol, investigators are examining the ability for a novel multiplex PCR assay with mixed floral antibiotic resistance profiling is safe and increases effective treatment for urinary tract infections in a urology clinic over traditional culture methods alone and decreases retreatment rates in this population.

DETAILED DESCRIPTION:
The novel multiplex real-time PCR assay with mixed floral antibiotic resistance profiling offers a higher degree of sensitivity and specificity than conventional culture methods in the identification of UTI pathogens as determined by the previous prospective comparison study. Additionally, conventional methods are often inadequate in the case of polymicrobial infections. More accurate and timely pathogen identification allows for prompt and more targeted treatment with less reliance on empiric therapy and decreased rates of antibiotic therapy changes and retreatment. This leads to more favorable patient outcomes and decreases the development of resistant organisms.

ELIGIBILITY:
Inclusion Criteria:

* • Patient Informed Consent form completed

  * Male and Female Subjects may participate with no predetermined quotas or ratios for gender participation.
  * All patients must be ≥60 years old. For patients presenting with a diagnosis of interstitial cystitis, patients may be of any age.
  * Patients must be presenting for treatment of acute UTI, complicated UTI, persistent UTI, or recurrent UTI's.
  * Including prostatitis, pyelonephritis, and/or interstitial cystitis.
  * Data pertaining to the times at which the specimen samples are collected and stabilized needs to be documented.
  * Specimen samples obtained need to have a sufficient volume necessary to perform a urine culture and Guidance 4.0.

Exclusion Criteria:

* • Do not provide written informed Consent with HIPAA authorization form.

  * Taking antibiotics for any reason other than UTI at the time of enrollment
  * Patients with chronic (> 10 days) indwelling catheters
  * Self-catheterized patients
  * Patients with neobladders

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2511 (Actual)
Dates: Start 2018-07-17 (Actual); Primary Completion 2019-02-22 (Actual); Study Completion 2019-10-01 (Actual)

PRIMARY OUTCOMES:
Establish Safety: composite adverse event rate | 7 Days
  Demonstrate safety of Guidance 4.0 multiplex real-time PCR organism identification with mixed floral antibiotic resistance profiling guided treatment. Safety will be measured with a composite adverse event outcome of urosepsis, pyelonephritis, hospitalization, or the need to attend an urgent care center. The composite adverse event rate in the arm tested with Guidance 4.0 will be shown to be non-inferior to that in the arm tested with traditional urine culture. Superiority will also be tested.

SECONDARY OUTCOMES:
Number of Patients with Recurrent and Persistent Infections in Each Arm | 7 Days
  Demonstrate non-inferiority and possibly superiority of Guidance 4.0 over traditional urine C&S with respect to the percentage of recurrent and persistent infections. Persistent is remaining infection at day 7 and recurrent infection is a person that had a second infection within 30 days that was treated with antibiotics.
Time to Symptom Resolution in Each Arm | 7 days
  Demonstrate superiority of Guidance 4.0 over traditional urine C&S with respect to the time to symptom resolution as demonstrated by UTISA tool. Symptom resolution will be defined as an overall rating of no symptoms on the UTISA questionnaire.

OTHER OUTCOMES:
Physician Choice for Decision Making when Provided Both Results | 4 Months
  • To determine which test physicians, rely upon when given the results of both traditional urine C&S vs. Guidance 4.0.

CONTACTS AND LOCATIONS:
Overall Officials: Kirk Wojno, MD, Principal Investigator — Comprehensive Urology
Locations (1):
- Comprehensive Urology, Royal Oak, Michigan, United States